CLINICAL TRIAL: NCT00419809
Title: A Placebo Controlled Study to Evaluate the Safety and Tolerability of Repeat Doses of SB-681323 in Patients Receiving Methotrexate for Rheumatoid Arthritis.
Brief Title: SB-681323-Methotrexate Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RA1101607
Record Dates: First submitted 2007-01-05; First posted 2007-01-09 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-01

CONDITIONS: Arthritis, Rheumatoid
Keywords: methotrexate,; SB-681323,; p38 MAP Kinase Inhibitor,; liver function; Rheumatoid Arthritis,
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — dilmapimod

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SB-681323 oral tablets

SUMMARY:
SB-681323 is a p38 MAP-kinase inhibitor that has potential uses in inflammatory conditions such as RA. Previous p38 MAP-kinase inhibitors have been hindered in development by liver toxicity. Methotrexate (common treatment for RA patients) also has potential liver toxicity. This study was an enabling study to determine the safety of co-administration of the two compounds with respect to liver function

ELIGIBILITY:
Inclusion Criteria:

* Male or female. Females must be of non-child-bearing capacity
* BMI 19 - 30 kg/m2 (inclusive)
* Diagnosis of RA according to the revised 1987 criteria of the American College of Rheumatology (ACR)
* Negative urine drugs of abuse screen, breath alcohol tests, hepatitis B and C, and HIV tests.
* Liver function tests within normal limits
* Must be on a stable dose of methotrexate (2.5 - 25 mg/week) for >8 weeks prior to enrolment and which will not be changed during the course of this study.
* Must be on stable folate supplements for >8 weeks prior to enrolment with normal red cell folate levels at enrollment.

Exclusion Criteria:

* History of alcohol &/or drug abuse
* Abnormal ECGs at screening
* Liver disease, uncontrolled hypertension, diabetes mellitus, psoriasis, history of peptic ulcer disease
* The patient is using glucocorticoid at doses >10mg/day.
* The patient is using sulphasalazine at a dose >3g/day.
* The patient is using hydroxychloroquine at a dose >400mg/day.
* The patient is on treatment regimen of DMARDs other than MTX plus one or both of sulphasalazine and hydrochloroquine (e.g. leflunomide)
* The patient dose of NSAIDs, COX-2 inhibitors or glucocorticoids change at any time during 2 weeks prior to enrolment until the end of the clinical phase of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-05; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the values of liver function tests following dosing with methotrexate alone (Day 1) and methotrexate and SB-681323 or placebo (Day 15).

SECONDARY OUTCOMES:
The other comparisons of interest is the pharmacokinetics of methotrexate when dosed alone (Day 1) relative to when dosed with SB681323 (Day 15) pharmacodynamics (effect of SB-681323 on CRP & IL-6 at Days 1, 8 and 15.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Australia (2):
  - GSK Investigational Site, Randwick, Sydney, New South Wales
  - GSK Investigational Site, Adelaide